CLINICAL TRIAL: NCT01046461
Title: A Phase II Study to Evaluate the Efficacy and Tolerability of Ramosetron, Aprepitant and Dexamethasone (RAD) in Preventing Cisplatin-induced Nausea and Vomiting in Chemotherapy-naïve Patients With Solid Cancer
Brief Title: Ramosetron, Aprepitant and Dexamethasone (RAD) in Solid Cancer
Acronym: RAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RAD1.0
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Solid Tumour; Postoperative Nausea and Vomiting
Keywords: Ramosetron; aprepitant; dexamethasone; cancer; chemotherapy; antiemetics; cisplatin; nausea; vomiting; high dose cisplatin
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Neoplasms; Nausea; Vomiting | interventions — ramosetron; Aprepitant; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramosetron, Aprepitant, Dexamethasone (Experimental)
  Interventions: Drug: Ramosetron, Aprepitant, Dexamethasone

INTERVENTIONS:
Drug: Ramosetron, Aprepitant, Dexamethasone — Day 1:
  Aprepitant 125 mg PO, 1 hour before chemotherapy Ramosetron 0.6 mg IV, 30 min before chemotherapy Dexamethasone 12 mg PO, 30 min before chemotherapy
  Day 2 - 3:
  Aprepitant 80 mg PO. in the morning Dexamethasone 8 mg PO. in the morning
  Day 4 Dexamethasone 8 mg PO. in the morning
  Other Names: Nasea; Emend

SUMMARY:
Cisplatin is one of the most emetogenic drugs used in clinical practice and it could result in poor compliance with chemotherapy. The 5-HT3 receptor antagonists prevent vomiting in acute phase emesis after chemotherapy in 73 - 92% of cisplatin-treated patients when coadministered with steroids, but they appear to lack efficacy in the delayed phase emesis. Ramosetron, a new 5-HT3 receptor antagonists, has been shown to have equivalent efficacy and tolerability and a longer duration of effect than granisetron in preventing acute vomiting in patients undergoing cisplatin-containing chemotherapy. Acute phase emesis was prevented in 84.8% of patients receiving ramosetron plus dexamethasone, but the CR rate of total phase emesis was less than 60%.

Aprepitant is a selective, high-affinity NK1 receptor antagonist. Adding aprepitant to 5-HT3 receptor antagonists and steroid improve CR rate of not only chemotherapy induced acute emesis and but also delayed emesis by 11-14 and 20 percentage points, respectively.

But until now, there was no information that which 5-HT3 receptor antagonists is the best partner for aprepitant. Therefore, we initiated a prospective, open-label, phase II study to assess the efficacy and tolerability of a combination of ramosetron, aprepitant and dexamethasone (RAD) in the prevention of cisplatin based CINV in chemotherapy-naïve patients with solid cancer

DETAILED DESCRIPTION:
Cisplatin is one of the most emetogenic drugs used in clinical practice and it could result in poor compliance with chemotherapy. The 5-HT3 receptor antagonists prevent vomiting in acute phase emesis after chemotherapy in 73 - 92% of cisplatin-treated patients when coadministered with steroids, but they appear to lack efficacy in the delayed phase emesis. Ramosetron, a new 5-HT3 receptor antagonists, has been shown to have equivalent efficacy and tolerability and a longer duration of effect than granisetron in preventing acute vomiting in patients undergoing cisplatin-containing chemotherapy. Acute phase emesis was prevented in 84.8% of patients receiving ramosetron plus dexamethasone, but the CR rate of total phase emesis was less than 60%.

ELIGIBILITY:
Inclusion Criteria:

* 18 -75 years, both sex
* ECOG performance status 0-2
* Histologically proven solid cancer, chemotherapy-naïve patient
* Planed to receive cisplatin (≥ 50mg/m2) based, single day chemotherapy,
* No nausea or vomiting within 72 hours prior to chemotherapy
* Serum Cr < 2.5 mg/dl, or calculated CCr ≥ 50 ml/min
* Serum total bilirubin < 2 mg/dl, AST/ALT < 3 times the upper normal limit , ALP < 5 times the upper normal limit
* Absolute neutrophil count ≥ 1,500/μL, platelet ≥ 100,000/μL
* Expected life duration ≥ 3 months
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, active gastric or duodenal ulcers, or pregnancy or breast-feeding
* Patients who should take steroid, antiemetics, pimozide, terfenadine, astemizole, cisapride, rifampin, carbamazepine, phenytoin, ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir or nelfinavir for the treatment of other diseases
* Patients taking any medicine, which could affect study results, within 1 week before chemotherapy (or taking anti-emetics within 48 hours before chemotherapy). Prior to beginning chemotherapy, single-agent benzodiazepines as hypnotic is allowed, but it can't be receiving during day 1-6 of 1st chemotherapy cycle.
* Patients with symptomatic brain metastasis
* Patients with GI obstruction or other diseases that could provoke nausea and vomiting
* Patients receiving RT on brain, abdomen or pelvis within 2 weeks before chemotherapy
* Patients who cannot understand informed consent or express his/her condition
* Patients who cannot swallow drugs
* Patients who have known allergy or severe side effect on study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate of RAD for the prevention of chemotherapy induced nausea vomiting (CINV) during overall phase (form 1 to 5 days) (overall phase is defined as acute and delayed phase) | from chemotherapy day 1 to day 5

SECONDARY OUTCOMES:
CR rate of RAD for the prevention of acute and delayed phase of CINV (from 0 to 24 hours /from 2 to 5 days) | until 1 month after chemotherapy
Severity of nausea | until 1 month after chemotherapy
Time to first occurrence of vomiting | until 1 month after chemotherapy
Adverse events reported using CTCAE v3.0 | until 1 month after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jung Kim, M.D., Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do, South Korea